CLINICAL TRIAL: NCT01533753
Title: Randomized, Open-Label Quality of Life Study Using Gabapentin Versus Venlafaxine in Treating Hot Flashes in Patients With Prostate Cancer
Brief Title: Quality of Life Study Using Gabapentin Versus Venlafaxine in Treating Hot Flashes in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO11813; 2011-0492 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); NCI-2012-00050 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2014-09

CONDITIONS: Prostate Cancer
Keywords: hot flashes; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes | interventions — Gabapentin; Venlafaxine Hydrochloride

ARMS (2):
- Arm A: Gabapentin (Experimental): Gabapentin will be administered orally at a starting dose of 300mg at bedtime (titration encouraged to desired effect and tolerability per treating physician). Maximum dose allowed will be 300mg three times a day. One cycle is defined as 28 +/- 7 days.
  Interventions: Drug: Gabapentin
- Arm B: Venlafaxine (Experimental): Venlafaxine will be administered orally at the starting dose of 37.5mg daily (titration allowed to desired effect and tolerability per treating physician). Maximum dose allowed will be 75mg per day. One cycle is defined as 28 +/- 7 days.
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Gabapentin — Gabapentin will be administered orally at a starting dose of 300mg at bedtime (titration encouraged to desired effect and tolerability per treating physician). Maximum dose allowed will be 300mg three times a day. One cycle is defined as 28 +/- 7 days.
  Other Names: Fanatrex; Gabarone; Gralise; Horizant; Neurontin
  Arms: Arm A: Gabapentin
Drug: Venlafaxine — Venlafaxine will be administered orally at the starting dose of 37.5mg daily (titration allowed to desired effect and tolerability per treating physician). Maximum dose allowed will be 75mg per day. One cycle is defined as 28 +/- 7 days.
  Other Names: Effexor
  Arms: Arm B: Venlafaxine

SUMMARY:
The purpose of this study is to assess the change in quality of life over a 6 month period between gabapentin and venlafaxine in men with prostate cancer treated for hot flashes related to androgen deprivation therapy.

DETAILED DESCRIPTION:
60 evaluable patients with prostate cancer currently receiving androgen ablation therapy or who have had an orchiectomy will be enrolled in this study. All patients will be randomized 1:1 (30 patients per treatment arm) to either receive gabapentin or venlafaxine. Treatment duration will be a total of 6 months. During those 6 months, study staff will evaluate frequency and intensity of hot flashes using hot flash score from hot flash diary every 28 days. Patients will also record side effects associated with either gabapentin or venlafaxine on their medication diaries. Study staff will record the severity of all adverse events reported. Patients will also complete the quality of life Functional Assessment of Cancer Therapy-Prostate (FACT-P) form at baseline, cycle 3, and cycle 6/off study.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years or older with histologically proven adenocarcinoma of the prostate
* Prior or current androgen deprivation for at least 6 months prior to study entry with either bilateral orchiectomy or being maintained on a stable dose of LHRH (luteinizing hormone-releasing hormone) agonist or antagonist

  * Hot flash frequency of an average of 2 or more per day (average of 14 hot flash episodes per week)

Exclusion Criteria:

* cannot currently be taking serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs) or monoamine oxidase inhibitors (MAOIs)

  * cannot have uncontrolled hypertension
  * cannot have history of past or current of epilepsy, epilepsy syndrome or other seizure disorder
  * cannot have psychiatric history of mania, hypomania, bipolar disorder or anorexia nervosa
  * cannot be receiving concurrent treatment with amy medications or herbal products being used with the express purpose of treating hot flashes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bruce, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics (Carbone Cancer Center), Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from medical clinic between the dates of 1/31/2012 and 5/9/2014.
Period: Overall Study
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1 | 3 | 4
  African American | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in Quality of Life
Description: We will measure the absolute change in the Functional Assessment of Cancer Therapy-Prostate (FACT-P) total score, between gabapentin and venlafaxine in men with prostate cancer treated for hot flashes related to androgen deprivation therapy
Time Frame: observed over a 6 month treatment period
Population: Zero participants analyzed due to early termination of study.
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare Toxicity Rates Between the Gabapentin and Venlafaxine Treatment Groups
Description: Toxicity rates will be compared between the two groups
Time Frame: over a 6 month treatment period
Population: Zero participants analyzed due to early termination of study
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Assess Changes in the Hot Flash Scores for the Two Arms
Description: Assess percentage changes in the hot flash score from baseline to cycle 6 between gabapentin and venlafaxine in men with prostate cancer treated with for hot flashes related to androgen deprivation therapy
Time Frame: 6 month treatment period
Population: Zero participants analyzed due to early termination of study
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Assess Changes in Quality of Life Using the Hot Flash Related Daily Interference Scale (HFRDIS)
Description: Assess percent change in quality of life from baseline to cycle 6, as measured by the Hot Flash Related Daily Interference Scale (HFRDIS) total score, between gabapentin and venlafaxine in men with prostate cancer treated for hot flashes related to androgen deprivation therapy.
Time Frame: over the 6 month treatment period
Population: Zero participants analyzed due to early termination of study
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of first dose of treatment through 6 months of treatment
Arm/Group | Arm A: Gabapentin | Arm B: Venlafaxine
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Gabapentin (N=2) | Arm B: Venlafaxine (N=3)
Systolic Ejection Murmur (Cardiac disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 1 (1)
Balance problem (Nervous system disorders) | 1 (1) | 0 (0)
Vivid Dreams (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to slow accrual. The data was uninterpretable due to the small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes